CLINICAL TRIAL: NCT03273452
Title: Chidamide With PET Regimen for Angioimmunoblastic T Cell Lymphoma, a Multicentric, Single Arm, Open Label Phase II Clinical Trial
Brief Title: Chidamide With PET Regimen for Angioimmunoblastic T Cell Lymphoma (PET: Prednisone, Etoposide and Thalidomide)
Acronym: PET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Principal Investigator, Hongwei Xue, MD., Qingdao University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Xuehw001
Record Dates: First submitted 2017-08-31; First posted 2017-09-06 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Angioimmunoblastic T-cell Lymphoma
MeSH Terms: conditions — Immunoblastic Lymphadenopathy | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Intervention Model Description: single arm trial, patients enrolled would be treated in this arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): In this group, patients will be given prednisone 100mg,qd,d1-5; etoposide 100mg,qd,d1-5; thalidomide 100mg,qn,d1-14; Chidamide 30mg,biw;
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — Chidamide will be given orally 30mg,biw, along with PET regimen (prednisone 100mg,po,qd,d1-5; etoposide 100mg,po,qd,d1-5; thalidomide 100mg,po,qn,d1-14;)
  Other Names: PCT regimen

SUMMARY:
This study aims to investigate the efficacy and safety of PET regimen combined with Chidamide for angioimmunoblastic T cell lymphoma patients.

DETAILED DESCRIPTION:
Patients enrolled in the trial would be given prednisone, etoposide, thalidomide and Chidamide, and the response and side effects are observed and documented.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed as angioimmunoblastic T cell lymphoma (diagnosed by pathologic department in IIIA hospitals or verified by certified institutions), immunohistochemistry should include: CD3, CD4, CD8, CD20, CD10, CD21, CD35, Bcl6, CXCL13, EBER, PD-1, Ki67.
2. At least on measurable focus (≥1.0*1.0cm by imaging), or at least one evaluable focus;
3. Age 18-75 years, both male and female;
4. ECOG 0-2, KPS≥ 70points;
5. Expected survival ≥3 months;
6. Peripheral blood neutrophil count ≥1.5×10^9/L, platelet count≥ 75×10^9/L, Hb≥ 90g/L;
7. Liver function: bilirubin ≤1.5 times of the normal maximum; AST、ALT≤2 times of the normal maximum (for patients with liver infiltration AST、ALT≤3 times of the normal maximum); renal function: blood creatinine ≤2 times the normal maximum;
8. Negative random pregnancy test for fertile women patients within 7 days before enrollment;
9. No radiation therapy, chemotherapy, targeted therapy nor hemopoietic stem cell transplantation within 4 weeks before enrollment;
10. No anti-tumor therapy at enrollment, including herbal therapy, immunotherapy and biologic therapy, symptomatic treatment is not within this range;

Exclusion Criteria:

1. Women during pregnancy or lactation, and fertile women that are not willing to take contraceptive measurements;
2. Patients with other malignant tumors simultaneously that have not been effectively controlled;
3. Patients with history of using HDAC inhibitors;
4. Patients who are allergic to medicine used in the trial, or have metabolic disorders toward these medicine;
5. Patients with severe active infection;
6. Patients with HIV or syphilis infection;
7. Patients with prolonged QT interval (male > 450ms，female > 470ms), or chronic heart failure patients with level III or IV cardiac function; or those have the following heart disease within 6 months before enrollment: acute coronary syndrome, acute heart failure (heart function level III or IV), distinctive ventricular arrhythmias (prolonged ventricular tachycardia, ventricular fibrillation, etc);
8. Patients with history of organ transplantation;
9. Patients with history of thrombosis and embolism;
10. Patients with mental disorders or those who are unable to sign a written consent;
11. Patients with drug abuse or long-time alcoholism that may influence the result of the trial;
12. Patients who do not have capacity of legal transactions;
13. Patients currently in other clinical trials;
14. Those who are recognized as inappropriate for the trial by the investigators;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate(ORR) | every 3 months until 24 months after the last patient's enrollment
  the rate of patients who achieve objective remission after the treatment,including CR (complete remission),CRu (complete remission with unrecovered platelet count) and PR (partial remission).

SECONDARY OUTCOMES:
duration of remission | from the day of remission to the date of first documented progression，up to 24 months after the last patient's enrollment
  from date of complete remission to date of progression, relapse, or death from any cause
progression free survival | from the day of treatment to the date of first documented progression，up to 24 months after the last patient's enrollment
  from date of inclusion to date of progression, relapse, or death from any cause
overall survival | 24 months after the last patient's enrollment
  from the date of inclusion to date of death, irrespective of cause

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
After the trial is finished, all the data would be available at the principle investigator's location.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Wang Y, Zhang M, Song W, Cai Q, Zhang L, Sun X, Zou L, Zhang H, Wang L, Xue H. Chidamide plus prednisone, etoposide, and thalidomide for untreated angioimmunoblastic T-cell lymphoma in a Chinese population: A multicenter phase II trial. Am J Hematol. 2022 May;97(5):623-629. doi: 10.1002/ajh.26499. Epub 2022 Mar 11. PMID 35170082